CLINICAL TRIAL: NCT01486940
Title: A Multi-centre, Multinational, Open-labelled, Randomised, Parallel-Group Comparison of Insulin Detemir Plus Insulin Aspart With NPH Insulin Plus Human Soluble Insulin in Subjects With Type 1 Diabetes on a Basal-Bolus Regimen
Brief Title: Comparison of Insulin Detemir Plus Insulin Aspart With Insulin NPH Plus Human Soluble Insulin in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1374
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin Aspart; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Basal/bolus regimen 1 (Experimental)
  Interventions: Drug: insulin detemir; Drug: insulin aspart
- Basal/bolus regimen 2 (Active Comparator)
  Interventions: Drug: insulin NPH; Drug: human soluble insulin

INTERVENTIONS:
Drug: insulin detemir — Individually adjusted dose administered subcutaneously (s.c., under the skin) twice daily
  Arms: Basal/bolus regimen 1
Drug: insulin aspart — Individually adjusted dose administered subcutaneously (s.c., under the skin) prior to meals
  Arms: Basal/bolus regimen 1
Drug: insulin NPH — Individually adjusted dose administered subcutaneously (s.c., under the skin) twice daily
  Arms: Basal/bolus regimen 2
Drug: human soluble insulin — Individually adjusted dose administered subcutaneously (s.c., under the skin) prior to meals
  Arms: Basal/bolus regimen 2

SUMMARY:
This trial is conducted in Europe and South America. The aim of this trial is to compare the glycaemic control of insulin detemir plus insulin aspart with that of insulin NPH plus human soluble insulin in subjects with type 1 diabetes on a basal/bolus regimen.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 12 months
* Current treatment with any basal/bolus regimen or any biphasic insulin treatment for at least 6 months
* BMI below or equal to 35 kg/m^2
* HbA1c below or equal to 12%

Exclusion Criteria:

* Proliferative retinopathy or maculopathy requiring acute treatment
* Recurrent major hypoglycaemia that may interfere with trial participation (as judged by the Investigator)
* Subjects with known hypoglycaemic unawareness as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2002-03; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin)

SECONDARY OUTCOMES:
Intra-subject variation in home measured blood glucose (3-point blood glucose profiles)
8-point blood glucose profiles
Incidence of self-recorded hypoglycaemic episodes
Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (65):
- Argentina (2):
  - Novo Nordisk Investigational Site, Junín
  - Novo Nordisk Investigational Site, Morón
- Novo Nordisk Investigational Site, Varaždin, Croatia
- Czechia (4):
  - Novo Nordisk Investigational Site, Hradec Králové
  - Novo Nordisk Investigational Site, Liberec
  - Novo Nordisk Investigational Site, Plzen - Lochotin
  - Novo Nordisk Investigational Site, Prague
- Denmark (9):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Copenhagen
  - Novo Nordisk Investigational Site, Hillerød
  - Novo Nordisk Investigational Site, Hjørring
  - Novo Nordisk Investigational Site, Holbæk
  - Novo Nordisk Investigational Site, Køge
  - Novo Nordisk Investigational Site, Silkeborg
  - Novo Nordisk Investigational Site, Slagelse
  - Novo Nordisk Investigational Site, Svendborg
- Finland (7):
  - Novo Nordisk Investigational Site, Kemi
  - Novo Nordisk Investigational Site, Kokkola
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Pärnu
  - Novo Nordisk Investigational Site, Rovaniemi
  - Novo Nordisk Investigational Site, Viljandi
- France (9):
  - Novo Nordisk Investigational Site, Angers
  - Novo Nordisk Investigational Site, Grenoble
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Lorient
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Mougins
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Poitiers
- Novo Nordisk Investigational Site, Athens, Greece
- Italy (13):
  - Novo Nordisk Investigational Site, Alessandria
  - Novo Nordisk Investigational Site, Asti
  - Novo Nordisk Investigational Site, Bari
  - Novo Nordisk Investigational Site, Bergamo
  - Novo Nordisk Investigational Site, Catania
  - Novo Nordisk Investigational Site, Genova
  - Novo Nordisk Investigational Site, Lucca
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Padua
  - Novo Nordisk Investigational Site, Prato
  - Novo Nordisk Investigational Site, Ravenna
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Torino
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Norway (7):
  - Novo Nordisk Investigational Site, Arendal
  - Novo Nordisk Investigational Site, Gjettum
  - Novo Nordisk Investigational Site, Gjøvik
  - Novo Nordisk Investigational Site, Kongsberg
  - Novo Nordisk Investigational Site, Kongsvinger
  - Novo Nordisk Investigational Site, Kristiansand
  - Novo Nordisk Investigational Site, Rådal
- Poland (6):
  - Novo Nordisk Investigational Site, Bydgoszcz
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Szczecin
- Novo Nordisk Investigational Site, Timișoara, Romania
- Novo Nordisk Investigational Site, Moscow, Russia
- Slovakia (2):
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Moldava nad Bodvou
- Novo Nordisk Investigational Site, Falun, Sweden

REFERENCES:
- [Result] Hermansen K, Fontaine P, Kukolja KK, Peterkova V, Leth G, Gall MA. Insulin analogues (insulin detemir and insulin aspart) versus traditional human insulins (NPH insulin and regular human insulin) in basal-bolus therapy for patients with type 1 diabetes. Diabetologia. 2004 Apr;47(4):622-9. doi: 10.1007/s00125-004-1365-z. PMID 15298338
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com